CLINICAL TRIAL: NCT00990509
Title: Albumin for Intracerebral Hemorrhage Intervention
Acronym: ACHIEVE
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Enrollment was stopped due to low recruitment and the PI's move to a different institution.
Sponsor: Georgetown University (Other)
Collaborators: Baxter Healthcare Corporation (Industry)
Responsible Party: Principal Investigator, Chelsea Kidwell, M.D., Professor of Neurology; Medical Director, Georgetown University Stroke Center, Georgetown University
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 2009-173
Record Dates: First submitted 2009-10-01; First posted 2009-10-07 (Estimated); Results first posted 2014-08-29 (Estimated); Last update posted 2014-08-29 (Estimated); Status verified 2014-08

CONDITIONS: Intracerebral Hemorrhage
Keywords: Primary ICH; Albumin; MRI; Neuroimaging outcome; Placebo-controlled; Phase II; Blinded; Safety; Acute ICH; ICH; Primary acute (< 48 hours) supratentorial ICH
MeSH Terms: conditions — Cerebral Hemorrhage | interventions — Albumins; Contrast Media

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Albumin (Experimental)
  Interventions: Drug: Albumin; Procedure: Brain MRI with and without contrast
- Placebo (Placebo Comparator)
  Interventions: Drug: Placebo; Procedure: Brain MRI with and without contrast

INTERVENTIONS:
Drug: Albumin — Three (3) daily IV infusions of 1.25 g/kg Albumin (25%) on Days 1-3 following enrollment.
  Other Names: BUMINATE 25%, Albumin (Human)
  Arms: Albumin
Drug: Placebo — Three (3) daily IV infusions of 1.25 g/kg Saline solution on Days 1-3 following enrollment
  Arms: Placebo
Procedure: Brain MRI with and without contrast — All subjects will receive 3 brain MRI studies, regardless of if they are randomized into Albumin or Placebo condition.
  MRIs will be with and without contrast will be performed at:
  * Baseline
  * 48 hours after enrollment(approximately Day 3)
  * 96 hours after drug treatment begins (approximately Day 5)
  Other Names: 1.5T Siemens Symphony MRI.; 3T Siemens Verio

SUMMARY:
The purpose of this study is to find out what effects, good and bad, the medication Albumin has on subjects who have experienced a type of stroke known as an intracerebral hemorrhage (ICH). An ICH is when spontaneous bleeding into the brain occurs due to fragile blood vessels.

This research is being done because currently there is no effective treatment for ICH. However, study investigators believe that Albumin, the medication being tested in this study, is safe and may help improve patient recovery from ICH over time.

Subjects will be enrolled in the study for a total of 90 days. Following enrollment, subjects will be randomized to receive 3 daily injections of either Albumin or Placebo (liquid with no drug), and will receive 3 brain MRI scans (with and without contrast), as described below.

All subjects will be monitored continuously through 96 hours after enrollment (5 days) in the Georgetown ICU. Blood tests and clinical evaluations of neurological status, consisting of questions about subjects' functional abilities and medical history, will occur in the Georgetown ICU once every 24 hours through post-enrollment Day 5. Additionally, subjects will receive daily chest x-rays, and daily EKGs (exams that monitor how your heart is doing by placing electrodes, or small monitors, on your skin in specific locations).

Similar clinical evaluations will occur at Day 30 and Day 90. Should subjects be discharged at these time points, day 30 assessments will occur over the phone, and day 90 assessments will occur in-person at Georgetown University Medical Center.

DETAILED DESCRIPTION:
We aim to determine the safety and explore the efficacy of human albumin as a neuroprotective (or cytoprotective) agent for the treatment of acute primary supratentorial ICH. Albumin therapy has been shown to be cytoprotective in animal studies of both ischemic stroke and intracerebral hemorrhage, and in a phase II human study in ischemic stroke.

To date no acute intervention (beyond supportive medical care) has been identified to improve outcomes in patients with primary ICH. Neuronal injury from a primary ICH is due not only to the space occupying effects of the hemorrhage but also due to the development of edema and toxicity from blood breakdown products in the subacute phase. Cytoprotective strategies targeted to limit blood brain barrier (BBB) breakdown and edema formation hold promise as treatment strategies to limit this injury.

A number of MR imaging outcome markers demonstrating a potential neuroprotective effect include measures of hematoma volume, perihematomal edema, and blood brain barrier disruption. The term "hyperintense acute injury marker" (HARM) has been proposed to describe the radiologic finding of hyperintense signal within the cerebrospinal fluid spaces visualized on post-contrast fluid attenuated inversion recovery (FLAIR) MRI in patients with acute ischemic stroke. HARM has the potential to serve as a marker of blood brain barrier disruption in patients with primary ICH. The current study will involve serial MR imaging in ICH patients randomized to placebo vs. albumin to assess whether there are differences in the frequency of HARM and perihematomal edema in the albumin treated patients.

ELIGIBILITY:
Inclusion Criteria:

* Primary supratentorial ICH
* < 48 hours from symptom onset
* Age >18
* Signed informed consent obtained from the patient or patient's legally authorized representative

Exclusion Criteria:

* ICH volume < 5 cc
* Glasgow Coma Scale < 6
* Surgical evacuation anticipated
* Pre-existing medical, neurological or psychiatric disease that would confound the neurological, functional, or imaging evaluations
* Pregnancy or breastfeeding
* Hemodynamic instability (SBP < 100 mmHg, > 200 mmHg)
* Current participation in another experimental treatment protocol
* Renal impairment with GFR < 30 or Creatinine > 2.0
* History of or known allergy to albumin
* History of or known severe allergy to rubber latex
* Episode/exacerbation of congestive heart failure (CHF) from any cause in the last 6 months. (An episode of congestive heart failure is any heart failure that required a change in medication, diet or hospitalization)
* Acute myocardial infarction in the last 6 months
* Elevated serum troponin level on admission > 0.1 mcg/L
* Known valvular heart disease with CHF in the last 6 months
* Known (or in the investigator's judgment) existence of severe aortic stenosis or mitral stenosis
* Cardiac surgery involving thoracotomy (e.g., coronary artery bypass graft (CABG), valve replacement surgery) in the last 6 months
* Suspicion of aortic dissection on admission
* Acute arrhythmia (including any tachy- or bradycardia) with hemodynamic instability on admission (systolic blood pressure < 100 mmHg).
* Findings on physical examination of any of the following: (1) jugular venous distention (JVP > 4 cm above the sternal angle); (2) 3rd heart sound; (3) resting tachycardia (heart rate > 100/min) attributable to congestive heart failure; (4) abnormal hepatojugular reflux; (5) lower extremity pitting edema attributable to congestive heart failure or without apparent cause; (6) bilateral rales; and/or (7) if a chest x-ray is performed, definite evidence of pulmonary edema, bilateral pleural effusion, or pulmonary vascular redistribution.
* Current acute or chronic lung disease requiring supplemental chronic or intermittent oxygen therapy.
* Prosthetic heart valves
* Contraindication to MRI (metal implant, etc.)
* Documented left ventricular ejection fraction < 35%

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 14 (Actual)
Dates: Start 2009-09; Primary Completion 2013-06 (Actual); Study Completion 2013-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Chelsea Kidwell, MD, Principal Investigator — Georgetown University
Locations (1):
- Georgetown University Hospital, Washington D.C., District of Columbia, United States

RESULTS

PARTICIPANT FLOW:
Groups:
- Albumin: Albumin: Three (3) daily IV infusions of 1.25 g/kg Albumin (25%) on Days 1-3 following enrollment.
  Brain MRI with and without contrast: All subjects will receive 3 brain MRI studies, regardless of if they are randomized into Albumin or Placebo condition.
  MRIs will be with and without contrast will be performed at:
  * Baseline
  * 48 hours after enrollment(approximately Day 3)
  * 96 hours after drug treatment begins (approximately Day 5)
- Placebo: Placebo: Three (3) daily IV infusions of 1.25 g/kg Saline solution on Days 1-3 following enrollment
  Brain MRI with and without contrast: All subjects will receive 3 brain MRI studies, regardless of if they are randomized into Albumin or Placebo condition.
  MRIs will be with and without contrast will be performed at:
  * Baseline
  * 48 hours after enrollment(approximately Day 3)
  * 96 hours after drug treatment begins (approximately Day 5)
Period: Overall Study
Arm/Group | Albumin | Placebo
Started | 5 | 9
Completed | 5 | 8
Not Completed | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Albumin | Placebo | Total
Number analyzed (Participants) | 5 | 9 | 14
Age, Continuous [Mean (Full Range); unit: years] | 62.6 [41 to 82] | 58.1 [41 to 76] | 59.7 [41 to 82]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 | 3 | 3
  Male | 5 | 6 | 11
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 1 | 1
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 3 | 5 | 8
  White | 2 | 3 | 5
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 0
  Not Hispanic or Latino | 5 | 9 | 14
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 5 | 9 | 14

OUTCOME MEASURES:

1. Primary Outcome: Mean Hyperintense Acute injuRy Marker (HARM)
Description: Hyperintense Acute injuRy Marker (HARM) characterizes the frequency and severity of blood brain barrier disruption. Mean HARM is assessed on the post-contrast study using a previously developed 5 point scale (0 to 5).). A score of 0 indicates no HARM, whereas a score of 5 indicates diffuse and generalized HARM. 11 of 14 participants received a Day 5 MRI. HARM reads could only be performed on 4 of the 7 placebo subjects due to insufficient sequences or presence of subarachnoid blood. Mean HARM score is presented.
Time Frame: Day 5 MRI
Measure: Number; unit: points
Arm/Group | Albumin | Placebo
Number analyzed (Participants) | 0 | 4
points |  | NA — Insufficient number of patients with outcome measure available for meaningful analysis as trial was stopped early. Analysis of a small number of observations would be misleading.

2. Primary Outcome: Assessment of Safety of Albumin Administration in Primary ICH
Description: Serious adverse events. Specific safety outcomes assessed: frank pulmonary edema as visualized on chest X-Ray, congestive heart failure, neurological deterioration (4-point worsening on NIHSS), death
Time Frame: Through Day 90 following enrollment
Measure: Number; unit: events
Arm/Group | Albumin | Placebo
Number analyzed (Participants) | 5 | 9
events
  Serious Adverse Events | 4 | 2
  Pulmonary Edema | 2 | 0
  Congestive Heart Failure | 0 | 0
  Neurological Deterioration | 1 | 0
  Death | 1 | 2

3. Primary Outcome: Mean Intracerebral Hemorrhage (ICH) Volume
Description: 11 of 14 participants received a Day 5 MRI. Mean ICH volume based on 11 participants is presented.
Time Frame: Day 5 MRI
Measure: Mean (Standard Deviation); unit: cc
Arm/Group | Albumin | Placebo
Number analyzed (Participants) | 4 | 7
cc | 41.2 (47.9) | 39.2 (31.5)

ADVERSE EVENTS:
Time Frame: 90 Days
Description: We did not collect non-serious adverse events.
Arm/Group | Albumin | Placebo
Serious Adverse Events (participants affected / at risk) | 4/5 | 2/9
Other Adverse Events (participants affected / at risk) | 0/0 | 0/0
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Albumin (N=5) | Placebo (N=9)
Pulmonary Edema (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 0 (0)
Neurologic Deterioration (Nervous system disorders) | 1 (1) | 0 (0) — The single event of neurologic deterioration documented in this study resulted in death due to respiratory failure and was adjudicated to be unrelated to the study interventions.
Death (General disorders) | 1 (1) | 2 (2)

LIMITATIONS AND CAVEATS:
There was an insufficient number of subjects in each treatment arm to allow for a meaningful analysis of the effects of albumin on HARM status (blood brain barrier disruption).

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No